#### STUDY PROTOCOL AND STATISTICAL ANALYSIS PLAN

#### Title:

Comparative Effects of High-Intensity Interval Training Modalities on Physical Performance and Physiological Responses in Competitive Table Tennis Players

#### **Brief Title:**

HIIT Effects on Table Tennis Players

### **Unique Protocol ID:**

E-77192459-050.99-376986

### **ClinicalTrials.gov Identifier:**

NCT Number: Not yet assigned

## **Document Type:**

Study Protocol and Statistical Analysis Plan

#### **Sponsor:**

Karabük University

### **Principal Investigator:**

Dr. Alirıza Han Civan

#### **Ethics Approval:**

Karabük University Non-Interventional Clinical Research Ethics Committee

**Decision No: 2024/1956** 

**Approval Number**: E-77192459-050.99-376986

**Approval Date: 27 September 2024** 

#### **Document Date:**

03 January 2026

### **Study Objectives**

To examine the comparative effects of calisthenic/plyometric HIIT and kettlebell-based Tabata HIIT on physical performance and physiological responses in competitive table tennis players.

### **Study Design**

Randomized, parallel-group experimental study conducted over 8 weeks.

# **Participants**

• Sample size: 24 male competitive table tennis players

• Age range: 18–24 years

- Inclusion criteria: actively training competitive athletes
- Exclusion criteria: musculoskeletal injury, cardiovascular or metabolic disease

#### **Interventions**

## **Group 1 – Calisthenic/Plyometric HIIT**

- Tabata-based HIIT protocol
- 3 sessions/week for 8 weeks
- Performed in addition to regular table tennis training

## **Group 2 – Kettlebell HIIT**

- Tabata-based HIIT protocol
- 3 sessions/week for 8 weeks
- Performed in addition to regular table tennis training

### **Outcome Measures**

## **Primary Outcomes:**

- Agility
- Flexibility
- Vertical jump
- VO<sub>2</sub>max

## **Secondary Outcomes:**

- Sprint performance
- Peak power
- Average power

#### **Data Collection**

Outcome measures assessed at baseline (pre-intervention) and post-intervention (8 weeks).

# **Statistical Analysis Plan**

• Software: SPSS and/or R

• Analysis population: Intention-to-treat

• Descriptive statistics: Mean  $\pm$  standard deviation

• Inferential analysis

## 2 × 2 mixed-design ANOVA

Within-subject factor: time (pre vs post)

Between-subject factor: group

Post-hoc paired-sample t-tests with Bonferroni correction

Statistical significance: p < 0.05

# Confidentiality

All participant data are anonymized. No identifying information is included in this document.

### INFORMED CONSENT FORM

### Title:

Comparative Effects of High-Intensity Interval Training Modalities on Physical Performance and Physiological Responses in Competitive Table Tennis Players

### **Unique Protocol ID:**

E-77192459-050.99-376986

## **ClinicalTrials.gov Identifier:**

NCT Number: Not yet assigned

## **Document Type:**

Informed Consent Form

#### **Sponsor:**

Karabük University

## **Principal Investigator:**

Dr. Alirıza Han Civan

#### Date:

27 September 2024

- Purpose of the study explained
- Procedures and exercises described
- Risks and potential benefits outlined
- Voluntary participation and right to withdraw stated
- Confidentiality and anonymization assured
- Contact information provided
- Signature lines for participant and investigator included